CLINICAL TRIAL: NCT05679492
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, add-on Phase III Clinical Study on the Efficacy and Safety of Meplazumab for Injection in Adults With Mild and Moderate COVID-19 Infections
Brief Title: Study on the Safety and Efficacy of Meplazumab for Injection Patients COVID-19
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Based on current epidemic situation in China, there is few Mild and Moderate COVID-19 patients.
Sponsor: Jiangsu Pacific Meinuoke Bio Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPZ-III-01
Record Dates: First submitted 2023-01-10; First posted 2023-01-11 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meplazumab (Experimental): First dose: 0.2 mg/kg - Day 1; second dose: 0.2 mg/kg - Day 8
  Interventions: Biological: Meplazumab foe injection
- Placebo (Placebo Comparator): First dose: control - Day 1; second dose: control - Day 8
  Interventions: Other: Normal saline

INTERVENTIONS:
Biological: Meplazumab foe injection — Meplazumab is a humanized anti-CD147 immunoglobulin 2 (IgG2) monoclonal antibody which is expected to block the binding of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) spike protein to the human host-cell-expressed CD147, thereby blocking entry of SARS-CoV-2 into human tissue. This expectation is based on in vitro functional studies using Vero E6 cells infected with SARS-CoV-2 that demonstrated effective meplazumab mediated virus gene copy number inhibition upwards of 90% as evaluated by quantitative polymerase chain reaction. Meplazumab may also inhibit COVID-19 associated cytokine storm syndrome based on inhibition of the pro inflammatory factor Cyclophilin A host-cell CD147 interaction.
  Arms: Meplazumab
Other: Normal saline — Normal saline
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, add-on Phase III clinical study.

Based on the "Diagnosis and Treatment Protocol for COVID-19 Pneumonia (Trial 10th edition)" and according to the results of phase I and Phase II clinical studies, one dose group and one placebo group were used in this experiment. The experimental group was add-on experimental drugs for basic treatment and the control group was add-on placebo for basic treatment. The clinical study was led by the First Affiliated Hospital of the Chinese People's Liberation Army, and 1320 adult subjects with mild and medium COVID-19 infection were enrolled in the First Affiliated Hospital of the Chinese People's Liberation Army, the Second Affiliated Hospital of the Chinese People's Liberation Army, the Special Medical Center of the Air Force, and the Third People's Hospital of Shenzhen. A ratio of 1 to 1 was randomly assigned to the experimental or placebo groups.Subjects should have tested positive for COVID-19 nucleic acid in a laboratory and developed at least one symptom of SARS-CoV-2 within 96 hours prior to medication. The administration schedule was on day 1 of the trial (intravenous infusion of Meplazumab or placebo once in the morning of D0; The dosage was 0.2 mg/kg. If the 12 common clinical symptoms of SARS-CoV-2 infection are not relieved.the first administration of D7, an additional dose of 0.2 mg/kg is given based on the body weight of the subjects.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, add-on Phase III clinical study.

Based on the "Diagnosis and Treatment Protocol for COVID-19 Pneumonia (Trial 10th edition)" and according to the results of phase I and Phase II clinical studies, one dose group and one placebo group were used in this experiment. The experimental group was add-on experimental drugs for basic treatment and the control group was add-on placebo for basic treatment. The clinical study was led by the First Affiliated Hospital of the Chinese People's Liberation Army, and 1320 adult subjects with mild and medium COVID-19 infection were enrolled in the First Affiliated Hospital of the Chinese People's Liberation Army, the Second Affiliated Hospital of the Chinese People's Liberation Army, the Special Medical Center of the Air Force, and the Third People's Hospital of Shenzhen. A ratio of 1 to 1 was randomly assigned to the experimental or placebo groups.Subjects should have tested positive for COVID-19 nucleic acid in a laboratory and developed at least one symptom of SARS-CoV-2 within 96 hours prior to medication. The administration schedule was on day 1 of the trial (intravenous infusion of Meplazumab or placebo once in the morning of D0; The dosage was 0.2 mg/kg. If the 12 common clinical symptoms of SARS-CoV-2 infection are not relieved (remission is defined as: the comprehensive score of the 12 common clinical symptoms of SARS-CoV-2 infection is reduced by at least 1 grade), after the first administration of D7, an additional dose of 0.2 mg/kg is given based on the body weight of the subjects.During hospitalization, each subject completed the relevant examination indicators of each visit according to the test requirements. The subjects can be discharged if they meet one of the following conditions: ① The discharge criteria of Diagnosis and Treatment Protocol for COVID-19 Infection (Trial 10th edition) (the condition is significantly improved, vital signs are stable, body temperature is normal for more than 24 hours, lung imaging lesion is significantly improved) and the nucleic acid test of COVID-19 is negative for 1 time; ② to the 14th day after the first administration; Before discharge, subjects should complete all discharge examinations, and after discharge, subjects do not need to do other examinations, but 12 common clinical symptoms of SARS-CoV-2 infection should be recorded every day until the symptoms return to normal (score: 0), and continue for at least 2 days. Long-term follow-up evaluation was conducted at D15-21 and D22-27 after administration by telephone to determine the safety of the test drug.On day 28 after the first dose (D28±2), subjects returned to the study center again for all group exit examinations. If the subject terminates the trial early for any reason, laboratory testing and chest imaging evaluation are required to complete the efficacy and safety assessment. During the trial, subjects were given.

Both the experimental group and the control group received basic treatment, including symptomatic drugs for 12 common clinical symptoms of SARS-CoV-2 infection. Because NSaids, glucocorticoids and antiviral drugs have great influence on the evaluation of experimental drugs, the following restrictions are made: 1. Subjects are not allowed to self-administer NSaids during the study if their fever is ≥38.5℃ and/or pain related symptoms are assessed as severe among the 12 common clinical symptoms of SARS-CoV-2 infection (score: 3 points), loxoprofen sodium 60 mg/ time, not more than 2 times during the test, and the specific medication information was truthfully recorded; 2. When the subject's symptoms are further aggravated and require loxoprofen sodium for more than 3 times or glucocorticoid drugs, Antiviral therapy (such as Paxlovid (Nematvir tablet/Ritonavir tablet combination package), azivudine tablets, Monoravir capsules, ambavir mab/Romisivir injection, human immunoglobulin for COVID-19 or convalescent plasma for convalescent patients), and other antipyretic and analgesic agents other than loxoprofen sodium prescribed in the protocol, The subjects were required to leave the group and complete the last follow-up before leaving the group.

During the study, the researcher can add examination items according to the actual situation, and all abnormal and clinically significant changes occurred in the subjects during the observation period and before leaving the group shall be followed up until the subjects return to normal or are deemed to be clinically insignificant by the researcher.

Study end is defined as the last visit of the last subject or the last data point used for statistical analysis, whichever is the latest. The last subject refers to the last enrolled case.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 80 (including 18 and 80 years old), male or female
2. The subject tested positive for SARS-CoV-2 by nucleic acid test within 96 hours (4 days) prior to initial administration
3. The patient is confirmed to be infected with the COVID-19, meeting the diagnostic criteria for mild or moderate patients in the latest version of the COVID-19 Pneumonia Diagnosis and Treatment Protocol (Trial 10th Edition) issued by the Chinese Health Commission, and has at least one symptom of SARS-CoV-2, such as fever, cough, shortness of breath, sore throat, diarrhea, vomiting and taste disturbance within 96 hours before the first administration of the drug
4. According to the 12 common symptom assessment forms of SARS-CoV-2 infection, the total symptom assessment score of the subjects before randomization was ≥ 2 points
5. There is at least one possible risk factor for severe/critical SARS-CoV-2: ① Age > 60 years old; (2) Patients with cardiovascular and cerebrovascular diseases (including hypertension), diabetes, chronic pulmonary diseases (chronic obstructive pulmonary disease, moderate to severe asthma), chronic liver and kidney diseases, tumors and other underlying diseases, and the disease should be in a stable period; (3) Immune dysfunction (such as AIDS patients, long-term use of corticosteroids or other immunosuppressive drugs to cause immune dysfunction); ④ Obesity (body mass index ≥30); ⑤ Heavy smokers; ⑥ Those who have not received SARS-CoV-2 vaccine
6. Agree to take highly effective contraceptive measures within 3 months after taking the experimental drug
7. The subject can communicate well with the researcher, understand and comply with the requirements of the study, and understand and sign the informed consent

Exclusion Criteria:

* (1) Severe patients with SARS-CoV-2 meet any of the following criteria

  1. Shortness of breath, breathing rate ≥ 30 times /min
  2. At rest, oxygen saturation (SpO2) ≤ 93% during air intake
  3. Progressive exacerbation of clinical symptoms, lung imaging showed obvious progression of lesions within 24 ~ 48 hours >50%

  (2) Critically ill patients with SARS-CoV-2 meet any of the following criteria
  1. Respiratory failure occurs and requires mechanical ventilation
  2. Shock occurs
  3. Combined with other organ failure requires ICU care (3) Allergic constitution, known allergic to the test drug and its components (4) Suspected or confirmed severe, active bacterial, fungal, viral, or other infections (other than COVID-19) that researchers believe may pose a risk when implementing interventions (5) Patients who underwent surgery or chemotherapy or radiotherapy within 28days prior to screening (6) The investigator considers that participation in the study should be prevented from any serious concomitant systemic disease, condition, or disorder (7) Any of the following drugs or treatments were used before screening:

  <!-- -->

  1. Antiviral therapy (e.g., Paxlovid (nematavir/ritonavir packaged in combination), azvudine tablets, monogravir capsules, ambavirumab/romissuvir injection, or for the duration of the study) is planned to be used within 3 half-life periods before the first dose. COVID-19 human immunoglobulin or convalescent plasma), glucocorticoids, IL-6 inhibitors, non-steroidal anti-inflammatory drugs (nsaids), antineoplastic drugs, anti-transplant rejection drugs, or immunomodulatory biologics
  2. Those who plan to receive vaccines (including but not limited to COVID-19 vaccine) within 28 days prior to screening or during the study period
  3. He is on dialysis (8) When screening, any of the laboratory test indicators meet the following standards

  <!-- -->

  1. ALT or AST >3ULN
  2. Total bilirubin ≥2 ULN
  3. White blood cell count > ULN
  4. Neutrophil absolute value < 0.5×109/L
  5. Platelet count < 100×109/L
  6. eGFR <60mL /min/ 1.73m2 (calculated by CKD-EPI formula) (9) Weight ≤40 kg (10) Dizzy needle dizzy blood (11) Participated in other drug clinical trials within 3 months prior to screening (12) Pregnant or lactating women or pregnancy-positive women (13) Hepatitis B surface antigen, hepatitis C antibody, treponema pallidum antibody, and human immunodeficiency virus (HIV) antibody were positive for any one of the results (14) Patients inappropriate for participation for any other reasons at the investigator's discretion.

Note:The investigator should ensure that a subject meets all inclusion criteria and does not meet any exclusion criteria at screening.If the conditions of a subject are changed (including laboratory test results)and meet any exclusion criterion at any time from the screening to the first administration,the subject shall beexcluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
12 cases of SARS-CoV-2 infection reached the duration of clinical recovery | Day 28
  During the 28-day trial,12 cases of SARS-CoV-2 infection reached the duration of clinical recovery The 12 clinical symptoms of SARS-CoV-2 infection include:nasal congestion or runny nose, dry or sore throat, cough, fever (body temperature), headache, muscle or body pain, shortness of breath (difficulty breathing), weakness or fatigue, shivering or chills, nausea (feeling like vomiting), number of vomiting and number of diarrhea Continuous recovery of clinical symptoms Definition: All 12 common clinical symptoms/signs of SARS-CoV-2 returned to normal and lasted for at least 2 days. Patients with different 12 indicators above were evaluated according to the actual clinical symptoms, and those without clinical symptoms were evaluated with "0 score (none)".

SECONDARY OUTCOMES:
The time and proportion of SARS-CoV-2 nucleic acid to turn negative | Day 28
  The time and proportion of SARS-CoV-2 nucleic acid to turn negative during the 28-day trial
12clinical symptoms of SARS-CoV-2 infection reached the proportion of clinical sustained recovery | Day 28
  During the 28-day trial period,12clinical symptoms of SARS-CoV-2 infection reached the proportion of clinical sustained recovery
The proportion of light/medium to heavy/critical types | Day 28
  The proportion of light/medium to heavy/critical types during the 28-day trial period
Change from baseline in each of the 12 clinical symptom assessments of SARS-Cov-2 infection | Day 28
  Change from baseline in each of the 12 clinical symptom assessments of SARS-Cov-2 infection during the 28-day trial:The score of individual clinical symptoms was performed on a scale scoring of 0 to 3:0 was classified as "none", 1 as "mild", 2 as "moderate", and 3 as "severe"
The time and rate of improvement from baseline in lung imaging during the 28-day tria | Day 28
  Definition of improvement in lung imaging:During the study period,changes in lung imaging from baseline were defined as improvement if they met any of the following criteria:1)Reduction in lesion diameter;2)The number of lesions decreased;3)The number of lung lobes involved in the lesions decreased

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of the Air Force Medical University, Xi'an, China